CLINICAL TRIAL: NCT00005802
Title: Chemotherapy (CT) Followed by Donor Lymphocyte Infusion (DLI) Plus Interleukin 2 (IL-2) for Patients With Relapse Acute Myeloid or Lymphoid Leukemia After Allogeneic Hematopoietic Transplant
Brief Title: Chemotherapy Followed by Donor White Blood Cells Plus Interleukin-2 in Treating Patients With Acute Myeloid or Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1380.00; FHCRC-1380.00; NCI-H00-0057; CDR0000067777 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — aldesleukin; Filgrastim; Cytarabine; Etoposide; fludarabine phosphate; Methotrexate; Mitoxantrone; Hydrocortisone; Radiotherapy

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cytarabine
Drug: etoposide
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mitoxantrone hydrochloride
Drug: therapeutic hydrocortisone
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill leukemia cells. Treating donor white blood cells with interleukin-2 in the laboratory may help them kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of interleukin-2 when given after chemotherapy and donor white blood cells and to see how well they work in treating patients with acute myeloid leukemia or acute lymphoid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of interleukin-2 following donor lymphocyte infusion and chemotherapy in patients with relapsed acute myeloid or lymphoid leukemia after allogeneic peripheral blood stem cell transplantation.
* Determine the toxicity and efficacy of this regimen in these patients.

OUTLINE: This is a dose escalation study of interleukin-2 (IL-2). Patients are stratified according to disease status after chemotherapy (acute myeloid leukemia (AML) in complete remission (CR) vs acute lymphoid leukemia (ALL) or AML not in CR).

Patients receive one of three induction chemotherapy regimens, depending on type of leukemia, prior treatment, and response.

* Regimen 1: Patients receive high dose cytarabine IV over 2 hours twice a day on days 1, 3, and 5.
* Regimen 2: Patients receive mitoxantrone IV over 15 minutes and etoposide IV over 30 minutes on days 1-5.
* Regimen 3: Patients receive fludarabine IV over 30 minutes on days 1-5, cytarabine IV over 2 hours on days 1-4, and filgrastim (G-CSF) subcutaneously beginning on day 1 and continuing until blood counts recover.

Patients with extramedullary relapse receive local radiotherapy. Patients with ALL or CNS relapse receive intrathecal methotrexate with or without hydrocortisone and cytarabine.

Patients receive one donor lymphocyte infusion IV over 15-30 minutes within 28-60 days after starting chemotherapy. On the same day, IL-2 IV is administered over 24 hours for 5 days. After 2 days rest, IL-2 is again administered continuously for 10 days.

Cohorts of 5 patients receive escalating doses of IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 5 patients experience dose limiting toxicities. Up to 40 patients are treated at the MTD.

Patients are followed monthly for 3 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 11-15 patients per year will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Relapsed acute myeloid leukemia or acute lymphoid leukemia after allogeneic peripheral blood stem cell transplantation (PBSCT), documented by 1 of the following:

  * Morphologic relapse defined as 1 or more of the following:

    * Peripheral blasts in absence of growth factor therapy
    * Bone marrow blasts greater than 5% of nucleated cells
    * Extramedullary (CNS, testicular, or other sites)
  * Flow cytometric relapse defined as appearance in peripheral blood or bone marrow of cells with abnormal immunophenotype consistent with leukemia recurrence and noted at pretransplant
  * Cytogenetic relapse defined as:

    * Appearance in 1 or more metaphases from bone marrow or peripheral blood cells of nonconstitutional cytogenetic abnormality noted in at least 1 cytogenetic study performed prior to transplant OR
    * New abnormality known to be associated with leukemia
* Allogeneic PBSCT from related (HLA identical and 1 antigen mismatch) OR unrelated (match) donor

  * Must have achieved complete remission after PBSCT
* Current donor must be same as prior donor

  * Age 10 and over

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* SWOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No congestive heart failure requiring diuretics
* No uncontrolled arrhythmia

Pulmonary:

* No pulmonary dysfunction requiring oxygen therapy
* No pneumonia or severe obstruction
* FEV_1 at least 50% of predicted OR no greater than 50% decline from baseline
* No severe restrictive lung disease (total lung capacity less than 60% or 50% declined from baseline) not due to leukemia

Other:

* No sepsis, aspergillosis, or other active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent cyclosporine or tacrolimus during induction chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. D. Flowers, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Clark JA, Turner ML, Howard L, Stanescu H, Kleta R, Kopp JB. Description of familial keloids in five pedigrees: evidence for autosomal dominant inheritance and phenotypic heterogeneity. BMC Dermatol. 2009 Jul 28;9:8. doi: 10.1186/1471-5945-9-8. PMID 19638218